CLINICAL TRIAL: NCT00199706
Title: 7.2% NaCl in 6% Hydroxyethyl Starch Versus Placebo - Effect on Intracranial Pressure and Haemodynamics in Subarachnoidal Haemorrhage (SAH) Patients.
Brief Title: HyperHAES Versus Placebo - Effect on Intracranial Pressure in SAH Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2002-SAHA; S-01264
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2005-11

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Intracranial Pressure; Intracranial Hypertension; Hypertonic Solutions; Saline Solutions, Hypertonic
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Hypertension

INTERVENTIONS:
Drug: 7.2% NaCl in 6% hydroxyethyl starch solution

SUMMARY:
The purpose of this study is to determine whether 7.2% NaCl in 6% hydroxyethyl starch will lower intracranial pressure (ICP) in SAH-patients with normal or moderately elevated ICP in a placebo controlled study, and to describe the haemodynamic effects.

DETAILED DESCRIPTION:
In the acute phase after a SAH, many patients need intensive care treatment to control the development of fatally increased intracranial pressure. One type of treatment used is osmotherapy. Traditionally mannitol has been the preferred drug, but the use of hypertonic saline solutions has gained more and more acceptance. The immediate effect seems to be equivalent or better than with mannitol, and there seem to be less adverse effects, such as hypovolemia, acute renal failure, hyponatremia, and rebound increase of ICP.

Most clinical studies in patients with life-threatening increase in ICP are observational, and show a predictable effect of hypertonic saline. We wanted to strengthen our own findings from such a study by applying the same study model but with a placebo control group in patients with only moderately elevated ICP.

We also wanted to document the haemodynamic effects, measuring cardiac output, intrathorasic blood volume and extravascular lung water.

ELIGIBILITY:
Inclusion criteria:

* Subarachnoid Hemorrhage, source of bleeding radiologically or surgically secured
* Age > 18 years
* Mechanically ventilated
* Sedated
* Stable hemodynamics
* Stable intracranial pressure between 10 - 20 mmHg

Exclusion criteria:

- Serum sodium > 160 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-04; Study Completion 2004-10

PRIMARY OUTCOMES:
Changes in intracranial pressure (ICP) measured as area under the curve (AUC) during the 210 minutes trial period

SECONDARY OUTCOMES:
Changes in cerebral perfusion pressure (CPP) measured as AUC
changes in cardiac output
intrathorasic blood volume
extravascular lung water
serum sodium levels during the 210 minutes trial period

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Bentsen, MD, Principal Investigator — Oslo University Hospital